CLINICAL TRIAL: NCT06527534
Title: Exploring the Effects of Filgotinib, an Oral JAK-1 Selective Inhibitor, Proteomic Profile and Micro-RNA Expression in Peripheral Blood Mononuclear Cell (PBMC) of Patients With Active Rheumatoid Arthritis (RA)
Brief Title: Filgotinib Effect on Proteomic Profile and Micro-RNA Expression in Patients With Active Rheumatoid Arthritis (RA)
Acronym: FILRA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Giovanni Adami, Principal Investigator, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 215CET - FILRA
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
Keywords: RA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Filgotinib (Experimental): Filgotinib 200 mg qd
  Interventions: Drug: Filgotinib
- Adalimumab (Active Comparator): Adalimumab 40 mg q2wk
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Filgotinib — Patients will receive pills of Filgotinib 200 mg qd for 12 weeks
  Arms: Filgotinib
Drug: Adalimumab — Patients will receive subcutaneous injections of Adalimumab 40 mg q2wk for 12 weeks
  Arms: Adalimumab

SUMMARY:
Purpose:

The study aims to investigate how Filgotinib affects proteins and micro-RNA in the blood of patients with rheumatoid arthritis. This could help understand its impact on inflammation and bone health in these patients.

Study Design:

This is a single-center, prospective randomized study.

DETAILED DESCRIPTION:
Population:

The study will include 30 patients with active rheumatoid arthritis: 15 patients treated with Filgotinib. 15 patients treated with Adalimumab (used as a comparison group).

Procedures:

Participants will have blood samples taken at the start and then every 4 weeks up to 12 weeks. These samples will be used to analyze changes in proteins and micro-RNA. Participants will continue their regular rheumatoid arthritis treatment during the study.

Primary Objective:

To observe changes in the metabolic profile (proteins and micro-RNA) in patients treated with Filgotinib.

Secondary Objectives:

Compare the metabolic profile changes between Filgotinib and Adalimumab. Identify metabolic factors associated with early clinical response to Filgotinib.

Safety and Data Management:

Adverse events will be monitored and reported. Patient confidentiality will be maintained according to privacy laws.

Study Duration:

Recruitment: 16 weeks. Patient involvement: 12 weeks. Total study duration: 28 weeks.

ELIGIBILITY:
Inclusion criteria

* Rheumatoid arthritis (RA) according to ACR/EULAR 2010 criteria with active disease (Disease Activity Score 28-joints C-reactive protein [DAS28 CRP] >5.1 and/or Clinical Disease Activity Index [CDAI] >22)
* Age > 18, <65 years
* Patients for whom treatment with filgotinib or adalimumab might be planned

Exclusion criteria

* History of major cardiovascular events or stroke
* History of venous thromboembolism
* Active smokers or past smokers >10 pack/years
* History of fragility fractures or severe osteoporosis (T score at total hip or femoral neck or lumbar spine ≤3.5)
* Treatment with bone-active medications (estrogens, bisphosphonates, denosumab, teriparatide, romosozumab)
* Chronic treatment with moderate to high dose of glucocorticoids (≥7.5 mg/day of prednisone equivalent for more than 3 months prior to enrollment), short term (<3 months) will be accepted if tapered, as clinically feasible, to <7.5 mg/day before enrollment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
micro RNA (miRNA) | 12 weeks
  Fold increase in miRNA intensity measurements on the base-two logarithmic scale

SECONDARY OUTCOMES:
Proteomic profile | 12 weeks
  Fold increase in proteins intensity measurements on the base-two logarithmic scale
American College of Rheumatology 20% Improvement (ACR20) | 12 weeks
  Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement (ACR20) Response at Week 12
Health Assessment Questionnaire-Disability Index (HAQ-DI) | 12 weeks
  Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 12 (range 0.000 - 3.000, higher numbers are worse)
Disease Activity Score 28 joints measured with CRP (DAS28-CRP) | 12 weeks
  Change From Baseline in Disease Activity Score 28 joints measured with CRP (DAS28-CRP) at Weeks 12 (range 0.96 - 8.61, higher numbers are worse)
36-Item Short Form Survey (SF-36) | 12 weeks
  Change From Baseline in 36-Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Week 12 (range 0 - 100, lower numbers are worse)
Functional Assessment of Chronic Illness Therapy (FACIT) | 12 weeks
  Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 12 (range 0 - 52, lower numbers are worse)
American College of Rheumatology 50% Improvement (ACR50) | 12 weeks
  Percentage of Participants Who Achieved ACR 50% Improvement (ACR50) at Weeks 12
Tender Joint Count | 12 weeks
  Change From Baseline in Individual ACR Component: Tender Joint Count Based on 68 Joints (TJC68) at Weeks 12
Swollen Joint Count | 12 weeks
  Change From Baseline in Individual ACR Component: Swollen Joint Count Based on 66 Joints (SJC66) at Weeks 12
Subject's Global Assessment of Disease Activity (SGA) | 12 weeks
  Change From Baseline in Individual ACR Component: Subject's Global Assessment of Disease Activity (SGA) at Weeks 12 (range 0 - 10, higher numbers are worse)
Physician's Global Assessment of Disease Activity (PGA) | 12 weeks
  Change From Baseline in Individual ACR Component: Physician's Global Assessment of Disease Activity (PGA) at Weeks 12 (range 0 - 10, higher numbers are worse)
Pain on Numeric Rating Scale (NRS) | 12 weeks
  Change From Baseline in Individual ACR Component: Subject's Pain Assessment at Weeks 12 (range 0 - 10, higher numbers are worse)
Clinical Disease Activity Index (CDAI) | 12 weeks
  Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 12 (range 0 - 76, higher numbers are worse)
Simplified Disease Activity Index (SDAI) | 12 weeks
  Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 12 (range 0 - 91, higher numbers are worse)

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Section, University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: No